CLINICAL TRIAL: NCT02670798
Title: Implementation of a Thromboelastography Guided Transfusion Protocol in Pediatric Neuromuscular Scoliosis Surgery
Brief Title: Thromboelastography Transfusion Protocol for Pediatric Neuromuscular Scoliosis Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expiration of funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201506098
Record Dates: First submitted 2015-12-08; First posted 2016-02-02 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Neuromuscular Scoliosis
Keywords: neuromuscular; scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Standard of care hematologic management in the operating room
- Study (Experimental): Standard of care hematologic management plus additional monitoring with the intervention of Thromboelastography laboratory testing and use of a thromboelastography-guided transfusion protocol.
  Interventions: Procedure: Thromboelastography laboratory testing

INTERVENTIONS:
Procedure: Thromboelastography laboratory testing — Laboratory test that monitors clotting properties of blood
  Other Names: TEG
  Arms: Study

SUMMARY:
The long-term goal of this study is to optimize the perioperative care of pediatric spinal deformity patients, minimizing perioperative complications and increasing cost-effectiveness of perioperative hematologic management. The objective of the proposed study, which is the initial step in pursuit of this goal, is to evaluate the effectiveness of thromboelastography (TEG) to monitor coagulation pathways and direct blood product replacement in pediatric neuromuscular spinal deformity surgery. The central hypothesis of this study is that TEG will decrease exposure to allogeneic packed red blood cells (PRBC). The rationale is that proven effectiveness of TEG in neuromuscular deformity may change the standard of care for hematologic management in neuromuscular spinal deformity cases and additionally set the stage for a multicenter trial in idiopathic pediatric deformity.

DETAILED DESCRIPTION:
To achieve the aims of this study, the investigators will perform a randomized clinical trial comparing thromboelastography with standard intraoperative monitoring of coagulation pathways in pediatric neuromuscular deformity surgery. All patients will receive the standard of care hematological management, including intravenous tranexamic acid (50mg/kg loading bolus, 5mg/kg/hr infusion until wound closure) during surgery. Patients randomized to the TEG group will receive standard of care plus TEG tests at four time points: at the time of incision, at completion of surgical exposure, at completion of instrumentation, and upon arrival to the PACU. TEG results will be used to guide fluid replacement, in the form of platelets, fresh frozen plasma, cryoprecipitate, or more tranexamic acid according to previously published protocols9. Data collected will include standard preoperative demographic data: gender, age, body mass index, diagnosis; standard spinal deformity radiographic measurements; and surgical data including operative time, estimated blood loss, and blood product replacement. The international normalized ratio (INR) will be obtained at wound closure, along with a complete blood count, for both groups as per standard of care. Postoperative data points collected will include allogeneic packed red cell transfusion volume, drain output (all drains discontinued on postoperative day #3), time to normal feeding (either home feeding tube rate or normal per os diet), and time to discharge. Perioperative complications will be collected and categorized according to Glassman et al.

Cost data related to the hospital stay and care of any perioperative complications data will be recorded. These will include costs related to antibiotics, length of stay (including prolonged intensive care unit stay), and perioperative transfusion requirements. To approximate the costs related to transfusion, the investigators will include costs of acquisition, storage, and administration. Similar costs related to any other blood product administration will be collected and assigned as needed. The investigators anticipate that patient reported quality of life scores will be similar between groups. As this may not be the case, the investigators will collect quality adjusted life year (QALY) data through the ACEND survey. These data will be collected at the preoperative visit and at the 6, 12, and 24 month followup points.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are patients undergoing posterior spinal fusions of 10 or more segments with neuromuscular scoliosis, between the ages of 12 and 18 years old.

Exclusion Criteria:

* Exclusion criteria include Jehovah's witness status, known preoperative bleeding/coagulation abnormalities, preoperative use of anticoagulants (e.g. Coumadin, enoxaparin), or known blood dyscrasias.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss | Day of surgery
  Amount of blood lost during perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Kelly, MD, Principal Investigator — Associate Professor of Orthopedic Surgery
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No